CLINICAL TRIAL: NCT00415558
Title: Prospective, Multicenter, Un-Blinded, Single Arm, Clinical Study Using the Guidant Microwave Ablation System Comprised of the Flex 10 Ablation Probe and Microwave Generator for Patients With Symptomatic Paroxysmal Atrial Fibrillation
Brief Title: Prospective Clinical Study of the Guidant Microwave Ablation System for the Treatment of PAF in the MIS Procedure
Status: Terminated | Phase: Not Applicable | Type: Interventional
Why Stopped: Low enrollment
Sponsor: Maquet Cardiovascular (Industry)
Responsible Party: Maquet Cardiovascular, Maquet Cardiovascular
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: VR2049541
Record Dates: First submitted 2006-12-20; First posted 2006-12-25 (Estimated); Last update posted 2009-06-09 (Estimated); Status verified 2009-06

CONDITIONS: Atrial Fibrillation
Keywords: Atrial Fibrillation
MeSH Terms: conditions — Atrial Fibrillation

INTERVENTIONS:
Device: Microwave Ablation System

SUMMARY:
The purpose of this prospective, single-arm, un-blinded, multi-site clinical study is to assess the safety and efficacy of the Microwave Ablation System for the treatment of symptomatic paroxysmal atrial fibrillation (PAF) in the minimally invasive surgical (MIS) procedure in approximately 30 patients at 6 investigational sites in the United States.

DETAILED DESCRIPTION:
The study population for this study will be comprised of patients who have been diagnosed with symptomatic (PAF) for at least 6 months prior to study entry. Patients will be qualified for the study if they meet stringent inclusion/exclusion criteria, signing an informed consent and agreeing to return for followup visits at 1, 3, 6, 9 and 12 months. All study patients will receive microwave ablation to treat their symptomatic PAF. The Microwave Ablation System will be used during a MIS procedure on a beating heart in order to ablate a specified lesion pattern.

ELIGIBILITY:
Inclusion Criteria:

* Patient is greater than or = 18 years of age
* Patient has documented symptomatic paroxysmal atrial fibrillation (PAF) refractory to at least 1 antiarrhythmic (Class IA, IC, III) drug.
* Patient has episodes of symptomatic AF including, but not limited to, palpitations, lightheadedness, fatigue, dyspnea, and/or chest pain.
* A minimum of a 6-month history of symptomatic paroxysmal AF (documented by patient report in the medical record).
* A minimum of 2 discrete symptomatic paroxysmal AF episodes in the month prior to study entry. Paroxysmal AF rhythm must be documented by objective evidence (12-lead electrocardiogram [ECG], Holter monitor, event monitor, or other telemetry rhythm strip) with the presence of sinus rhythm and/or underlying rhythm between episodes.
* Patient has been informed of the nature of the study, agreed to its provisions, and provided written informed consent.

Exclusion Criteria:

* Patient had a cerebral vascular accident or transient ischemic attack within the previous 6 months.
* Patient had a myocardial infarction within the previous 6 weeks.
* Patient has underlying metabolic etiology related to AF (e.g., hyperthyroidism, metabolic disorder).
* Patient has significant underlying structural heart disease (e.g., valvular disease, presence of aneurysm, left ventricular hypertrophy) requiring surgical or procedural intervention.
* Patient with prior catheter ablation procedure for the treatment of AF within the previous 6 months.
* Patient has evidence of, or history of, 50% or more stenosis in any pulmonary vein.
* Patient had a previous thoracic procedure resulting in sternal opening and/or pericardial opening (e.g., surgical ablation, coronary artery bypass graft [CABG], or valve repair).
* Patient has a left atrial size > 6.0 cm measured on echocardiogram.
* Patient has a left ventricular ejection fraction (LVEF) < 35%.
* Patient requires treatment for CAD (coronary artery disease) or has untreated unstable angina.
* Patient has a presence of esophageal fistula or esophageal stricture, untreated esophagitis, varices, dysphagia, or odynophagia caused by anatomical abnormality or other diseases contraindicating transesophageal echocardiography.
* Patient has severe chronic obstructive pulmonary disease.
* Patient has a known allergy or contraindication to Coumadin (warfarin) therapy, or inability to comply with Coumadin (warfarin) therapy.
* Patient has a known allergy or contraindication to complying with antiarrhythmic (Class IA, IC, III) therapy.
* Patient has an acute illness or active systemic infection or sepsis.
* Patient has a co-morbidity with life expectancy of less than one year or protocol non-compliance that would limit follow-up.
* Patient is geographically remote and/or unable to return for follow-up examinations.
* Patient is pregnant or is planning to become pregnant during the study.
* Patient is enrolled in any concurrent study.

Min Age: 18 Years | Sex: All
Age Groups: Adult, Older Adult
Dates: Start 2007-05

CONTACTS AND LOCATIONS:
Overall Officials: Li Poa, MD, Principal Investigator — Enloe Medical Center; Dudley Hudspeth, MD, Principal Investigator — Banner Desert Medical Center; Daniel Bethencourt, MD, Principal Investigator — Long Beach Memorial Medical Center; Niloo Edwards, MD, Principal Investigator — University of Wisconsin Hospitals and Clinics; Norbert Baumgartner, MD, Principal Investigator — Covenant Medical Center
Locations (5):
- United States (5):
  - Mesa, Arizona
  - Chico, California
  - Long Beach, California
  - Saginaw, Michigan
  - Madison, Wisconsin